CLINICAL TRIAL: NCT07059676
Title: Design and Validation of Plasma Proteins and Cytokine Panels to Identify Markers Associated With Response to Niraparib as Maintenance Treatment After First-line Platinum-based Regimen in Patients With Advanced Ovarian Cancer
Acronym: LIBINI-1
Status: Not yet recruiting | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: LIBINI-1
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-05

CONDITIONS: Advanced Ovarian Cancer
MeSH Terms: interventions — niraparib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — liquid biopsy profiles of ovarian cancer patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Zejula (Niraparib): Profiles of ovarian cancer patients with sustained niraparib benefit as maintenance in the first line
  Interventions: Drug: Zejula (Niraparib)

INTERVENTIONS:
Drug: Zejula (Niraparib) — PARPi inhibitors have been incorporated into managing first-line advanced ovarian cancer with different approvals depending on homologous recombination (HR) status. Niraparib has received approval independent from HR status. Although the benefit is more remarkable in HR-deficient patients, there is no biomarker to predict sustained response to niraparib at the start of treatment helping the clinician to make decisions among the different treatment options.

SUMMARY:
PARPi inhibitors have been incorporated into managing first-line advanced ovarian cancer with different approvals depending on homologous recombination (HR) status. Niraparib has received approval independent from HR status. Although the benefit is more remarkable in HR-deficient patients, there is no biomarker to predict sustained response to niraparib at the start of treatment helping the clinician to make decisions among the different treatment options.

The aim of the LIBINI-1 (Liquid biopsy for predicting niraparib benefit if 1st line) study is to identify predictive biomarkers of sustained response to niraparib using liquid biopsy with two different technologies:

1. Proteomic and secretome analysis tools. The first part of the LIBINI-1 project is to create a platform for rapid screening and analysis by multiple detections of niraparib response-associated proteins in patients with advanced ovarian cancer.
2. ctDNA analysis. The second part of the LIBINI-1 project is to correlate the baseline level of ctDNA and change in ctDNA at 4 and 12 weeks with the benefit to niraparib.

DETAILED DESCRIPTION:
The main objective of this study (LIBINI-1 first part) is characterizing liquid biopsy profiles of ovarian cancer patients with sustained niraparib benefit as maintenance in the first line through proteomic and secretome analysis. The first part of LIBINI-1 is addressed by four individual subsequent objectives (see ANNEX 2).

Therefore, the primary objective is the development of a panel for multiplex detection of proteins associated with sustained benefit from niraparib maintenance.

For the execution of the primary objective the following consecutive secondary objectives are planned:

1. Global characterization of proteins (proteome) in plasma samples from patients with and without benefit from niraparib maintenance. Identification of molecular pathways of proteins differentially expressed between both groups.
2. Analysis of secreted proteins (secretome) in plasma samples of patients with and without benefit from niraparib maintenance.

3 & 4: Development of customized panels for multiplex detection of proteins associated with sustained benefit from niraparib maintenance.

After this discovery phase, the predictive panel should be validated in a confirmatory study with a larger cohort of advanced ovarian cancer patient samples.

The second part of LINIBI-1 is to correlate the baseline levels of ctDNA and the changes in ctDNA at 4 and 12 weeks (3 months) with benefit to niraparib. This second part of LIBINI-I will be analyzed in a subsequent study.

ELIGIBILITY:
Inclusion Criteria

1. Signed informed consent and ability to comply with treatment and follow up.
2. Patients ≥ 18 years old.
3. ECOG 0-1
4. Histologically confirmed diagnosis of FIGO stage III-IV high-grade serous or endometrioid ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
5. BRCA status according to local practice is known. It is encouraged to have BRCA testing in tumor.
6. Homologous recombination status according to local practice is encouraged.
7. Patients must meet the following front-line therapy requirements:

   1. Patients must have received at least 4 cycles of platinum-based therapy
   2. Patients must have non-evidence of disease or achieved a complete or partial response to platinum-based regimen Patient must meet all the required criteria for niraparib maintenance as single agent after first line platinum-based chemotherapy and receive niraparib therapy according to local prescribing information (see ANNEX 3).

Exclusion Criteria

1. According to niraparib's local prescribing information (see ANNEX 3): Patients must not be pregnant, breastfeeding, or expecting to conceive children while receiving study treatment and for 6 months after the last dose of study treatment. Women of childbearing potential must have a negative serum pregnancy test result within 72 hours prior to initiation of study treatment and have to use an effective contraceptive method along the participation in the study.
2. Patients must not have a known hypersensitivity to the components of niraparib or the excipients.
3. Patients must not have received prior treatment with a known PARP inhibitor.
4. Patients must not have had any known, persistent (>4 weeks), ≥Grade 3 hematological toxicity or fatigue from prior cancer therapy.
5. Patients must not have any known history of myelodysplastic syndrome (MDS) or a pretreatment cytogenetic testing result at risk for a diagnosis of MDS/acute myeloid leukemia (AML).
6. Patients must not have symptomatic uncontrolled brain or leptomeningeal metastases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: profiles of ovarian cancer patients with sustained niraparib benefit as maintenance in the first line
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Multiplex protein detection panel - Early progression | 0-24 months
  To identify a multiplex protein detection panel based on protein and cytokine from plasma at baseline and at 4 and 12 weeks from baseline, associated with early progression, defined as progression in the first 6 months after initiation of niraparib maintenance.
Multiplex protein detection panel - Absence of progression | 0-24 months
  To identify a multiplex protein detection panel based on protein and cytokine from plasma at baseline and at 4 and 12 weeks from baseline, associated with absence of progression at 18 months after initiation of niraparib maintenance

SECONDARY OUTCOMES:
Multiplex protein detection panel - Progression | 0-12 months
  To identify a multiplex protein detection panel based on protein and cytokine from plasma at baseline and at 4 and 12 weeks from baseline, associated to progression in the first 12 months after initiation of niraparib maintenance.
Multiplex protein detection panel - Absence of progression (12 + 24 months) | 0-24 months
  To identify a multiplex protein detection panel based on protein and cytokine from plasma at baseline and at 4 and 12 weeks from baseline, associated to absence of progression at 12 and 24 months after initiation of niraparib maintenance
Plasma protein identification - Progression | 0-12 months
  To identify proteins in plasma at baseline and at 4 and 12 weeks from baseline, associated to progression in the first 6 and 12 months after initiation of niraparib maintenance.
Plasma protein identification - Absence of progression | 0-24 months
  To identify proteins in plasma at baseline and at 4 and 12 weeks from baseline, associated to absence of progression at 12, 18 and 24 months after initiation of niraparib maintenance.
Plasma cytokines identification - Progression | 0-12 months
  To identify cytokines in plasma at baseline and at 4 and 12 weeks from baseline, associated to progression in the first 6 and 12 months after initiation of niraparib maintenance.
Plasma cytokines identification - Absence of progression | 0-24 months
  6. To identify cytokines in plasma at baseline and at 4 and 12 weeks from baseline, associated to absence of progression at 12, 18 and 24 months after initiation of niraparib maintenance.

IPD SHARING:
Plan to Share IPD: No